CLINICAL TRIAL: NCT00523848
Title: Phase II Study of VDT (VELCADE, Doxil® and Thalidomide) as Frontline Therapy for Patients With Previously Untreated Multiple Myeloma (MM)
Brief Title: Bortezomib, Doxorubicin Hydrochloride Liposome, and Thalidomide as First-line Therapy in Treating Patients With Previously Untreated Stage I, II, or III Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000563183; RPCI-I-59105 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2013-09-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Patients receive low-dose oral thalidomide once a day on days 1-28, bortezomib IV on days 1, 4, 15, and 18, and doxorubicin hydrochloride liposome IV over 60-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: bortezomib; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: thalidomide

INTERVENTIONS:
Drug: bortezomib — IV
Drug: pegylated liposomal doxorubicin hydrochloride — IV
Drug: thalidomide — Oral

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Giving bortezomib together with doxorubicin hydrochloride liposome and thalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with doxorubicin hydrochloride liposome and thalidomide works as first-line therapy in treating patients with previously untreated multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall response rate (complete response and partial response) in patients previously untreated stage I, II, or III multiple myeloma.

Secondary

* To evaluate the complete response rate in patients treated with this regimen.
* To determine the time to disease progression from the start of this therapy in patients treated with this regimen.

OUTLINE: Patients receive low-dose oral thalidomide once a day on days 1-28, bortezomib IV on days 1, 4, 15, and 18, and doxorubicin hydrochloride liposome IV over 60-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with residual disease who continue to show response after completion of 6 courses may receive 2 additional courses for a total of 8 courses.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I, II, or III multiple myeloma requiring therapy
* No prior systemic therapy for multiple myeloma

  * Patients who have received steroids or radiotherapy for cord compression or spinal cord disease are eligible for this study
  * Patients who have received 1 prior course of antimyeloma therapy may be enrolled at the investigator's discretion provided disease progression is not noted

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* Platelet count ≥ 75,000 cells/mm^3 (< 75,000 cells/mm^3 secondary to extensive bone marrow disease allowed at the PI's discretion with appropriate transfusion support)
* ANC ≥ 1,000 cells/mm^3
* Hemoglobin ≥ 8.0 g/dL (< 8 g/dL secondary to extensive bone marrow disease allowed at the PI's discretion with appropriate transfusion support)
* Creatinine clearance > 20 mL/min
* AST and ALT ≤ 2 times upper limit of normal (ULN) OR ≤ 3 times ULN (in the presence of liver metastases)
* Alkaline phosphatase ≤ 2 times ULN OR ≤ 3 times ULN (in the presence of liver metastases)
* Total bilirubin ≤ 2 times ULN OR ≤ 3 times ULN (in the presence of liver metastases)
* Ejection fraction ≥ 50% by MUGA or 2-D echocardiogram
* Negative pregnancy test
* Fertile patients must use at least 1 highly effective and 1 additional effective contraception method 4 weeks prior to, during, and 3 months after completion of study therapy
* HIV-negative
* Must have sufficient mental capacity to understand the explanation of the study and to provide informed consent
* Willingness and ability to comply with the FDA-mandated S.T.E.P.S. program

Exclusion criteria:

* Pregnant or lactating
* Active, serious infections uncontrolled by antibiotics
* Any medical condition or reason that, in the investigator's opinion, makes the patient unsuitable to participate in this clinical trial
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride or the components of doxorubicin hydrochloride liposome or bortezomib, boron, or mannitol
* Any of the following conditions:

  * History of uncontrolled New York Heart Association class II-IV heart disease or clinical evidence of congestive heart failure
  * Myocardial infarction within the past 6 months
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias, ECG evidence of acute ischemia, or active conduction system abnormalities
* Peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-06; Primary Completion 2011-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lee, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - VDT: VELCADE, Doxil and Low-dose Thalidomide: Patients receive low-dose oral thalidomide once a day on days 1-28, bortezomib IV on days 1, 4, 15, and 18, and doxorubicin hydrochloride liposome IV over 60-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm 1 - VDT: VELCADE, Doxil and Low-dose Thalidomide
Started | 46
Treated With Study Therapy | 44
Completed | 22
Not Completed | 24
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 2
Not completed — NOT TREATED (Became ineligible) | 2
Not completed — Disease Progression | 5
Not completed — Other, unspecified | 4

BASELINE CHARACTERISTICS:
Population: Evaluable Patients
Arm/Group | VDT: VELCADE, Doxil and Low-dose Thalidomide
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.13 (9.34)
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial)
Time Frame: Every 3 months
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VDT: VELCADE, Doxil and Low-dose Thalidomide
Number analyzed (Participants) | 40
percentage of participants | 77.50 [61.55 to 89.16]

2. Secondary Outcome: Complete Response Rate
Time Frame: Every 3 months
Population: Evaluable patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VDT: VELCADE, Doxil and Low-dose Thalidomide
Number analyzed (Participants) | 40
percentage of participants | 22.50 [10.84 to 38.45]

3. Secondary Outcome: Time to Disease Progression
Time Frame: Every 3 monthsntil the date of first documented progression or date of death from any cause, whichever came first
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | VDT: VELCADE, Doxil and Low-dose Thalidomide
Number analyzed (Participants) | 40
months | 27.8 [17.7 to 32.1]

ADVERSE EVENTS:
Arm/Group | VDT: VELCADE, Doxil and Low-dose Thalidomide
Serious Adverse Events (participants affected / at risk) | 16/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VDT: VELCADE, Doxil and Low-dose Thalidomide (N=44)
Febrile neutropenia - Grade 3 (Blood and lymphatic system disorders) | 1 (1)
Bradycardia - Grade 2 (Cardiac disorders) | 1 (1)
Cardiac failure congestive - Grade 3 (Cardiac disorders) | 2 (2)
Sinus bradycardia - Grade 2 (Cardiac disorders) | 1 (1)
Hypothyroidism - Grade 2 (Endocrine disorders) | 1 (1)
Asthenia - Grade 2 (General disorders) | 1 (1)
Chills - Grade 1 (General disorders) | 1 (1)
Oedema peripheral - Grade 3 (General disorders) | 1 (1)
Pain - Grade 2 (General disorders) | 2 (2)
Pyrexia - Grade 1 (General disorders) | 2 (2)
Pyrexia - Grade 2 (General disorders) | 1 (1)
Pyrexia - Grade 3 (General disorders) | 1 (1)
Pneumococcal bacteraemia - Grade 3 (Infections and infestations) | 1 (1)
Pneumonia - Grade 3 (Infections and infestations) | 6 (6)
Sepsis - Grade 3 (Infections and infestations) | 1 (1)
Lipids abnormal - Grade 1 (Investigations) | 1 (1)
Cachexia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Dehydration - Grade 2 (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Back pain - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache - Grade 1 (Nervous system disorders) | 1 (1)
Polyneuropathy - Grade 3 (Nervous system disorders) | 1 (1)
Spinal cord compression - Grade 3 (Nervous system disorders) | 1 (1)
Suicide attempt - Grade 4 (Psychiatric disorders) | 1 (1)
Renal failure acute - Grade 2 (Renal and urinary disorders) | 1 (1)
Dyspnoea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension - Grade 2 (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VDT: VELCADE, Doxil and Low-dose Thalidomide (N=44)
Anaemia - Grade 1 (Blood and lymphatic system disorders) | 8 (9)
Anaemia - Grade 2 (Blood and lymphatic system disorders) | 9 (9)
Anaemia - Grade 3 (Blood and lymphatic system disorders) | 2 (2)
Leukopenia - Grade 1 (Blood and lymphatic system disorders) | 19 (22)
Leukopenia - Grade 2 (Blood and lymphatic system disorders) | 11 (15)
Leukopenia - Grade 3 (Blood and lymphatic system disorders) | 7 (7)
Lymphopenia - Grade 1 (Blood and lymphatic system disorders) | 13 (14)
Lymphopenia - Grade 2 (Blood and lymphatic system disorders) | 14 (15)
Lymphopenia - Grade 3 (Blood and lymphatic system disorders) | 11 (11)
Neutropenia - Grade 1 (Blood and lymphatic system disorders) | 6 (7)
Neutropenia - Grade 2 (Blood and lymphatic system disorders) | 13 (16)
Neutropenia - Grade 3 (Blood and lymphatic system disorders) | 8 (9)
Neutropenia - Grade 4 (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia - Grade 1 (Blood and lymphatic system disorders) | 7 (11)
Thrombocytopenia - Grade 2 (Blood and lymphatic system disorders) | 4 (5)
Thrombocytopenia - Grade 3 (Blood and lymphatic system disorders) | 2 (2)
Bradycardia - Grade 1 (Cardiac disorders) | 3 (3)
Cyanosis - Grade 1 (Cardiac disorders) | 1 (1)
Tachycardia - Grade 1 (Cardiac disorders) | 1 (1)
Deafness - Grade 1 (Ear and labyrinth disorders) | 1 (1)
Deafness - Grade 2 (Ear and labyrinth disorders) | 1 (1)
Ear pain - Grade 1 (Ear and labyrinth disorders) | 1 (1)
Blepharitis - Grade 2 (Eye disorders) | 1 (1)
Diplopia - Grade 1 (Eye disorders) | 1 (1)
Dry eye - Grade 2 (Eye disorders) | 1 (1)
Eye swelling - Grade 1 (Eye disorders) | 1 (1)
Eyelid ptosis - Grade 2 (Eye disorders) | 1 (1)
Lacrimation increased - Grade 1 (Eye disorders) | 1 (1)
Meibomianitis - Grade 2 (Eye disorders) | 1 (1)
Vision blurred - Grade 1 (Eye disorders) | 4 (4)
Vision blurred - Grade 2 (Eye disorders) | 1 (1)
Visual disturbance - Grade 1 (Eye disorders) | 1 (1)
Abdominal discomfort - Grade 1 (Gastrointestinal disorders) | 1 (1)
Abdominal distension - Grade 1 (Gastrointestinal disorders) | 4 (4)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper - Grade 1 (Gastrointestinal disorders) | 1 (1)
Constipation - Grade 1 (Gastrointestinal disorders) | 27 (27)
Diarrhoea - Grade 1 (Gastrointestinal disorders) | 10 (12)
Dry mouth - Grade 1 (Gastrointestinal disorders) | 1 (1)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 3 (3)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Flatulence - Grade 1 (Gastrointestinal disorders) | 1 (1)
Haemorrhoids - Grade 1 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 1 (Gastrointestinal disorders) | 10 (11)
Stomatitis - Grade 1 (Gastrointestinal disorders) | 2 (2)
Vomiting - Grade 1 (Gastrointestinal disorders) | 6 (6)
Asthenia - Grade 1 (General disorders) | 8 (8)
Asthenia - Grade 2 (General disorders) | 1 (1)
Axillary pain - Grade 1 (General disorders) | 1 (1)
Chest discomfort - Grade 1 (General disorders) | 1 (1)
Chest pain - Grade 1 (General disorders) | 1 (1)
Chills - Grade 1 (General disorders) | 4 (4)
Fatigue - Grade 1 (General disorders) | 22 (24)
Fatigue - Grade 2 (General disorders) | 6 (7)
Fatigue - Grade 3 (General disorders) | 3 (3)
Feeling hot - Grade 1 (General disorders) | 1 (1)
Gait disturbance - Grade 1 (General disorders) | 3 (3)
Gait disturbance - Grade 2 (General disorders) | 1 (1)
Influenza like illness - Grade 1 (General disorders) | 3 (3)
Non-cardiac chest pain - Grade 1 (General disorders) | 2 (2)
Oedema - Grade 1 (General disorders) | 5 (5)
Oedema - Grade 2 (General disorders) | 1 (1)
Oedema peripheral - Grade 1 (General disorders) | 14 (15)
Oedema peripheral - Grade 2 (General disorders) | 2 (2)
Pain - Grade 1 (General disorders) | 4 (4)
Pain - Grade 2 (General disorders) | 1 (1)
Pyrexia - Grade 1 (General disorders) | 8 (8)
Tenderness - Grade 1 (General disorders) | 1 (1)
Xerosis - Grade 1 (General disorders) | 1 (1)
Hyperbilirubinaemia - Grade 1 (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia - Grade 2 (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity - Grade 1 (Immune system disorders) | 1 (1)
Hypersensitivity - Grade 1 (Immune system disorders) | 1 (1)
Bacterial infection - Grade 2 (Infections and infestations) | 1 (1)
Breast cellulitis - Grade 2 (Infections and infestations) | 1 (1)
Cystitis - Grade 1 (Infections and infestations) | 1 (1)
Eye infection - Grade 1 (Infections and infestations) | 1 (1)
Fungal infection - Grade 2 (Infections and infestations) | 1 (1)
Furuncle - Grade 2 (Infections and infestations) | 1 (1)
Hordeolum - Grade 1 (Infections and infestations) | 1 (1)
Infection - Grade 1 (Infections and infestations) | 2 (2)
Lobar pneumonia - Grade 2 (Infections and infestations) | 1 (1)
Localised infection - Grade 2 (Infections and infestations) | 1 (1)
Nasopharyngitis - Grade 1 (Infections and infestations) | 3 (3)
Oral candidiasis - Grade 1 (Infections and infestations) | 2 (2)
Oral candidiasis - Grade 2 (Infections and infestations) | 1 (2)
Pneumonia - Grade 1 (Infections and infestations) | 1 (1)
Pneumonia - Grade 2 (Infections and infestations) | 4 (5)
Pneumonia - Grade 3 (Infections and infestations) | 1 (1)
Rash pustular - Grade 1 (Infections and infestations) | 1 (1)
Sinusitis - Grade 1 (Infections and infestations) | 1 (1)
Tinea cruris - Grade 1 (Infections and infestations) | 1 (1)
Tinea infection - Grade 1 (Infections and infestations) | 1 (1)
Tinea pedis - Grade 2 (Infections and infestations) | 1 (1)
Upper respiratory tract infection - Grade 1 (Infections and infestations) | 1 (1)
Open wound - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased - Grade 1 (Investigations) | 5 (5)
Alanine aminotransferase increased - Grade 2 (Investigations) | 1 (1)
Aspartate aminotransferase increased - Grade 1 (Investigations) | 14 (14)
Aspartate aminotransferase increased - Grade 2 (Investigations) | 2 (2)
Blood alkaline phosphatase - Grade 1 (Investigations) | 2 (2)
Blood alkaline phosphatase increased - Grade 1 (Investigations) | 9 (11)
Blood creatine increased - Grade 1 (Investigations) | 3 (3)
Blood creatine increased - Grade 2 (Investigations) | 1 (1)
Heart rate decreased - Grade 1 (Investigations) | 1 (1)
Heart rate decreased - Grade 2 (Investigations) | 1 (1)
International normalised ratio increased - Grade 1 (Investigations) | 1 (1)
Weight decreased - Grade 1 (Investigations) | 1 (1)
Weight decreased - Grade 2 (Investigations) | 1 (1)
Weight decreased - Grade 3 (Investigations) | 1 (1)
Weight increased - Grade 1 (Investigations) | 1 (1)
Anorexia - Grade 1 (Metabolism and nutrition disorders) | 11 (11)
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Anorexia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite - Grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia - Grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia - Grade 1 (Metabolism and nutrition disorders) | 13 (13)
Hyperglycaemia - Grade 2 (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia - Grade 3 (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia - Grade 1 (Metabolism and nutrition disorders) | 9 (14)
Hyperkalaemia - Grade 2 (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia - Grade 1 (Metabolism and nutrition disorders) | 8 (11)
Hypernatraemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia - Grade 4 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 1 (Metabolism and nutrition disorders) | 4 (5)
Hypoalbuminaemia - Grade 2 (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia - Grade 1 (Metabolism and nutrition disorders) | 11 (11)
Hypocalcaemia - Grade 2 (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia - Grade 1 (Metabolism and nutrition disorders) | 8 (9)
Hypoglycaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia - Grade 1 (Metabolism and nutrition disorders) | 6 (9)
Hyponatraemia - Grade 1 (Metabolism and nutrition disorders) | 9 (10)
Hyponatraemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Oral intake reduced - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Arthralgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 6 (6)
Back pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain - Grade 3 (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness - Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal stiffness - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity - Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity - Grade 2 (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in jaw - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Amnesia - Grade 1 (Nervous system disorders) | 1 (1)
Balance disorder - Grade 1 (Nervous system disorders) | 1 (1)
Burning sensation - Grade 1 (Nervous system disorders) | 1 (1)
Cluster headache - Grade 1 (Nervous system disorders) | 1 (1)
Disturbance in attention - Grade 1 (Nervous system disorders) | 1 (1)
Dizziness - Grade 1 (Nervous system disorders) | 17 (22)
Dizziness - Grade 2 (Nervous system disorders) | 1 (1)
Dysgeusia - Grade 1 (Nervous system disorders) | 3 (3)
Dysgeusia - Grade 2 (Nervous system disorders) | 1 (1)
Headache - Grade 1 (Nervous system disorders) | 2 (3)
Hypoaesthesia - Grade 1 (Nervous system disorders) | 2 (3)
Hypoaesthesia - Grade 2 (Nervous system disorders) | 1 (1)
Neuropathy - Grade 1 (Nervous system disorders) | 3 (4)
Neuropathy - Grade 3 (Nervous system disorders) | 1 (1)
Neuropathy peripheral - Grade 1 (Nervous system disorders) | 11 (11)
Neuropathy peripheral - Grade 2 (Nervous system disorders) | 3 (3)
Neuropathy peripheral - Grade 3 (Nervous system disorders) | 1 (1)
Paraesthesia - Grade 1 (Nervous system disorders) | 4 (4)
Parosmia - Grade 1 (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy - Grade 1 (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy - Grade 1 (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy - Grade 2 (Nervous system disorders) | 1 (1)
Tremor - Grade 1 (Nervous system disorders) | 5 (5)
Anxiety - Grade 1 (Psychiatric disorders) | 1 (2)
Confusional state - Grade 2 (Psychiatric disorders) | 1 (1)
Confusional state - Grade 4 (Psychiatric disorders) | 1 (1)
Illusion - Grade 1 (Psychiatric disorders) | 1 (1)
Insomnia - Grade 1 (Psychiatric disorders) | 1 (1)
Nervousness - Grade 1 (Psychiatric disorders) | 1 (1)
Panic attack - Grade 1 (Psychiatric disorders) | 1 (1)
Sleep disorder - Grade 1 (Psychiatric disorders) | 1 (1)
Dysuria - Grade 1 (Renal and urinary disorders) | 1 (1)
Pollakiuria - Grade 1 (Renal and urinary disorders) | 1 (1)
Polyuria - Grade 1 (Renal and urinary disorders) | 1 (1)
Renal tubular acidosis - Grade 2 (Renal and urinary disorders) | 1 (1)
Pelvic pain - Grade 1 (Reproductive system and breast disorders) | 2 (2)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dysphonia - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Dyspnoea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccups - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal swelling - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Blister - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Decubitus ulcer - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Drug eruption - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin - Grade 1 (Skin and subcutaneous tissue disorders) | 10 (10)
Dry skin - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema - Grade 1 (Skin and subcutaneous tissue disorders) | 6 (6)
Erythema - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome - Grade 3 (Skin and subcutaneous tissue disorders) | 3 (3)
Pigmentation disorder - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 10 (11)
Rash - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Rash erythematous - Grade 1 (Skin and subcutaneous tissue disorders) | 6 (6)
Rash erythematous - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Rash erythematous - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash morbilliform - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin atrophy - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3)
Skin exfoliation - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis - Grade 3 (Vascular disorders) | 1 (1)
Hypertension - Grade 2 (Vascular disorders) | 1 (1)
Hypotension - Grade 1 (Vascular disorders) | 1 (1)
Hypotension - Grade 2 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 1 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 2 (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes